CLINICAL TRIAL: NCT00480077
Title: Diagnostic Outcome Trial in Heart Failure
Brief Title: Diagnostic Outcome Trial in Heart Failure (DOT-HF Trial)
Acronym: DOT-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment rates
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20061016-V2
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Heart Failure, randomized, OptiVol® Fluid status monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Intervention: in the access arm the patiens had programmmed the audible OptiVol Fliud status alert "on". Control patienst had programmed the audible alert "off"
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Access Arm (Experimental): HF subjects managed with standard clinical assessment and using the audible OptiVol® Fluid status monitoring alert and the device Cardiac Compass Report
  Interventions: Device: Programming (CRT-D, ICD OptiVol® and Cardiac Compass® )
- Control arm (Active Comparator): HF subjects managed with standard clinical assessment
  Interventions: Device: Programming (CRT-D, ICD OptiVol® and Cardiac Compass® )

INTERVENTIONS:
Device: Programming (CRT-D, ICD OptiVol® and Cardiac Compass® ) — OptiVol® Fluid status Monitoring with Cardiac Compass
  Other Names: OptiVol® audible alert

SUMMARY:
The DOT-HF trial is an international, prospective, multi-center, randomized, controlled trial.

DETAILED DESCRIPTION:
The study was designed with a Control Arm in order to adequately study the effect of early intervention triggered by the OptiVol® Alert and/or SentryCheck™ Monitor/PatientLook™ Indicator and evaluation using OptiVol® Fluid Status Monitoring with Cardiac Compass. OptiVol® Fluid Status Monitoring with Cardiac Compass features are available in the per Clinical Investigational Plan specified Medtronic products (CRT, CRT-D and ICD devices)

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders with mild to severe HF as defined as NHYA Class II to IV who also have an indication for device implant according to ESC/AHA guidelines as well as having a HF hospitalization or Emergency Department visit necessitating therapy within the past 12 months and who meet all inclusion criteria and no exclusion criteria, are eligible for this study.

Exclusion Criteria:

* Subject is post heart transplant or actively listed on the transplant list and reasonable probability (as defined by investigator) of undergoing transplantation in the next year
* Subject received a coronary artery bypass graft or valve surgery in last 90 days
* Subject with a myocardial infarction (MI) in the last 40 days.
* Subject's life expectancy is less than one year in the opinion of the physician
* Subject has severe Chronic Obstructive Pulmonary Disease (COPD), as determined by physician and documented in medical records
* Subject is listed for valve replacement/valve repair
* Subject has severe, primary pulmonary hypertension as determined by physician and documented in medical records
* Subject with serum creatinine ≥ 2.5 mg/dL measured within 14 days prior to enrolment
* Subject on chronic renal dialysis
* Subject on continuous or uninterrupted (≥ 2 stable infusions per week) infusion (inotropic) therapy for HF
* Subject has complex and uncorrected Congenital Heart Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2007-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. D.J. van Veldhuisen, MD, Study Chair — Groningen University Hospital, The Netherlands; Prof. Dr. med. M. Borggrefe, Study Chair — Ruprecht-Karls-Universität Heidelberg, Germany; Prof. Dr. V. Conraads, Principal Investigator — Universitair Ziekenhuis Brussel; Prof. C.M. Yu, Principal Investigator — Prince of Wales Hospital, Shatin, Hong Kong; Dr. F. Braunschweig, Principal Investigator — Karolinska University Hospital; Prof. Dr. J. Kautzner, Principal Investigator — IKEM- Klinika Kardiologie, Czech Republic; Prof. Dr. G. Jondeau, Principal Investigator — Hôpital Bichat Claude Bernard, France; Prof. Dr. M.R. Cowie, Principal Investigator — National Heart & Lung Institute, United Kingdom; Dr. R. Muñoz-Aguilera, Principal Investigator — Hospital General Universitario Gregorio Marañon, Spain; Prof. I. Ford, Principal Investigator — Robertson Center for Biostatistics, Scotland; Dr. M Lunati, Principal Investigator — Azienda Ospedaliera Niguarda Ca' Granda
Locations (1):
- Medtronic Bakken Research Center, Maastricht, Netherlands

REFERENCES:
- [Result] van Veldhuisen DJ, Braunschweig F, Conraads V, Ford I, Cowie MR, Jondeau G, Kautzner J, Aguilera RM, Lunati M, Yu CM, Gerritse B, Borggrefe M; DOT-HF Investigators. Intrathoracic impedance monitoring, audible patient alerts, and outcome in patients with heart failure. Circulation. 2011 Oct 18;124(16):1719-26. doi: 10.1161/CIRCULATIONAHA.111.043042. Epub 2011 Sep 19. PMID 21931078
- [Derived] Conraads VM, Spruit MA, Braunschweig F, Cowie MR, Tavazzi L, Borggrefe M, Hill MR, Jacobs S, Gerritse B, van Veldhuisen DJ. Physical activity measured with implanted devices predicts patient outcome in chronic heart failure. Circ Heart Fail. 2014 Mar 1;7(2):279-87. doi: 10.1161/CIRCHEARTFAILURE.113.000883. Epub 2014 Feb 11. PMID 24519908

RESULTS

PARTICIPANT FLOW:
Groups:
- Access Arm: HF subjects managed with standard clinical assessment and using OptiVol® Fluid status monitoring with Cardiac Compass Report
  Programming (CRT-D, ICD OptiVol® and Cardiac Compass® ) : OptiVol® Fluid status Monitoring with Cardiac Compass
- Control Arm: HF subjects managed with standard clinical assessment
  Programming (CRT-D, ICD OptiVol® and Cardiac Compass® ) : OptiVol® Fluid status Monitoring with Cardiac Compass
Period: Overall Study
Arm/Group | Access Arm | Control Arm
Started | 168 | 167
Completed | 137 | 141
Not Completed | 31 | 26
Not completed — Death | 19 | 15
Not completed — early exit | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Access Arm: HF subjects managed with standard clinical assessment and using OptiVol® Fluid status monitoring with Cardiac Compass Report
  Programming (CRT-D, ICD OptiVol® and Cardiac Compass® ): OptiVol® Fluid status Monitoring with Cardiac Compass
- Total: Total of all reporting groups
Arm/Group | Access Arm | Control Arm | Total
Number analyzed (Participants) | 168 | 167 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] — patient age and SD is similar between the 2 arms
  years | 64 (10) | 64 (10) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 146 | 142 | 288
QRS duration [Mean (Standard Deviation); unit: ms] | 142 (39) | 143 (36) | 142 (38)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28 (5) | 27 (4) | 28 (4)
NYHA functional class [Number; unit: participants] — Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  participants
    NYHA functional class I | 6 | 5 | 11
    NYHA functional class II | 98 | 103 | 201
    NYHA functional class III | 63 | 58 | 121
    NYHA functional class IV | 1 | 1 | 2
LVEF [Mean (Standard Deviation); unit: %] | 25 (7) | 25 (7) | 25 (7)
Type of device implanted [Count of Participants; unit: Participants]
  CRT-D | 141 | 133 | 274
  ICD | 27 | 34 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Combined End Point of All-cause Mortality or Heart Failure Hospitalization
Description: Number of participants with a combined end point of all-cause mortality or heart failure hospitalization
Time Frame: 14.9 ± 5.4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Access Arm | Control Arm
Number analyzed (Participants) | 168 | 167
Participants | 48 | 33
Statistical Analysis 1: Comparison: Access Arm vs Control Arm; Test type: Superiority — The primary end point of the study, all-cause death or hospitalization for heart failure, was analyzed on a time-to-first-event basis with the log-rank test. The hazard ratio (HR) associated with allocation to the access arm relative to control was estimated with corresponding 95% confidence interval (CI) by fitting a Cox proportional hazards model containing the treatment group as a categorical factor; p = 0.063, Log Rank

ADVERSE EVENTS:
Time Frame: mean follow up period (months): 14.9 +/- 5.4
Arm/Group | Access Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 50/168 | 34/167
Other Adverse Events (participants affected / at risk) | 47/168 | 20/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Access Arm (N=168) | Control Arm (N=167)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 39 (57) | 23 (32)
Pneumonia (Infections and infestations) | 6 (6) | 4 (5)
Lead Dislodgement (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Access Arm (N=168) | Control Arm (N=167)
Cardiac failure (Cardiac disorders) | 7 (10) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 7 (9) | 0 (0)
Chest pain (General disorders) | 8 (9) | 3 (3)
Oedema peripheral (General disorders) | 6 (8) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No